CLINICAL TRIAL: NCT04976673
Title: A Comparison of Clinical Efficiency of Photodynamic Therapy and Topical Corticosteroid in Treatment of Oral Lichen Planus- Split-Mouth Randomised
Brief Title: Comparison of Clinical Efficiency of Photodynamic Therapy and Topical Corticosteroid in Treatment of Oral Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: kb256/2020
Record Dates: First submitted 2021-06-15; First posted 2021-07-26 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-06

CONDITIONS: Lichen Planus, Oral
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Triamcinolone Acetonide; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Intervention Model Description: full contralateral split-mouth
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- photodynamic therapy side (Experimental): On one side, the OLP lesion eligible for treatment was subjected to photodynamic therapy in four sessions every 2 days.Using as photosensitizer Methylen blue for 10min the lesion was irradiated with a 650 nm semiconductor laser at a dose of 120 J / cm2
  Interventions: Procedure: Photodynamic Therapy
- Steroid side (Active Comparator): on the other side The OLP on the other side was treated by daily sticking a cut-to-size carrier with 0.05% triamcinolone acetonide for 8 days
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — The OLP on the other side was treated by daily sticking a cut-to-size carrier with 0.05% triamcinolone acetonide for 8 days
  Other Names: topical steroid administration
  Arms: Steroid side
Procedure: Photodynamic Therapy — the olp was photosensitized with methylen blue and was irradiated with a semiconductor laser with a wavelength of 650 nm, using a dose of 120 J / cm2 and power density
  Other Names: PDT
  Arms: photodynamic therapy side

SUMMARY:
Lichen planus is a chronic inflammatory dermatosis. It most often affects the skin and mucous membranes. Sometimes lesions may appear in the area of nails (estimated at 10% of patients) or genital organs and anus.

The most dangerous form of lichen planus is lichen that develops on the oral mucosa. It is believed to be the cause of the development of oral cancer.

The vast majority of people suffering from lichen planus - 90%, experience spontaneous resolution of symptoms within a maximum of two years from the moment of their onset.

In about half of the patients, the changes disappear within about 6 months. People who have a problem that their ailments do not want to go away on their own must take into account the fact that treating lichen is not the easiest one.

Treatment of lichen is mainly based on alleviating its symptoms and accelerating the resolution of symptoms. Topical ointments containing strong glucocorticosteroids are usually applied to skin lesions or we can use Photodynamic Therapy

DETAILED DESCRIPTION:
Oral lichen planus is most often characterized by lesions resembling a painless white mesh, which is usually located on the inside of the cheeks and the sides of the tongue. Lumps, erosions or erythematous changes are less often noticeable.

Symptoms in oral lichen planus are often:

reddening, dry mouth baking, swelling and minor bleeding.

Sometimes the gum mucosa exfoliates. When erosions occur, patients complain of pain and problems with drinking and swallowing food. Oral lesions necessarily require treatment.

Since lichen planus comes in many forms, some of them require histopathological examination to identify some of them. These tests involve taking a slice of the affected skin and examining it under a microscope.

Some causes of lichen planus are thought to involve several components.

Medications: lichen planus can occur as a reaction to certain medications, including:

beta-blockers, which are common drugs used to treat cardiovascular problems; anti-inflammatory drugs; injections to treat arthritis; antimalarial drugs; thiazide diuretics; phenothiazines, a group of tranquilizers with antipsychotic effects.

A prospective, randomized, single-blind 12-week clinical trial of full contralateral split-mouth in patients with bilateral erythematous or erosive lichen planus in the mouth.On one side, the OLP lesion eligible for treatment was subjected to photodynamic therapy using toluidine blue in four sessions every 2 days.

olp on the other side was treated with the administration of the steroid triamcinolone for 8 days

The clinical evaluation of the evolution of OLP eruptions was performed within 12 weeks of qualifying for treatment: at baseline, at the end of both treatments (day 8) and after the next 11 weeks

ELIGIBILITY:
Inclusion Criteria:

* having a histological diagnosis of OLP
* non smoker
* without diabetes melitus
* without hepatitis

Exclusion Criteria:

* diabetes melitus
* hepatitis
* occurrence dysplasia in the histopathological specimen;
* use of lichenoid reaction inducing medications and presence of amalgam fillings nearby the lesions;
* interventions for OLP in the previous 12 weeks;
* pregnant or breastfeeding women;
* proved or suspected hypersensitivity to any of the chemicals used in the treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-05-22 (Actual)

PRIMARY OUTCOMES:
Size of Oral lichen planus | 12 weeks
  the size of the oral lichen planus on oral mucosa in millimeters was assessed using a periodontal probe PCPUNC 15
  we measured the height and length of the lesions

SECONDARY OUTCOMES:
Pain rating | 12 weeks
  Pain ailments were assessed with the use of VAS (visual analog scale)
  Scale from 0 to 10 0 =no pain 10= maximal pain

CONTACTS AND LOCATIONS:
Overall Officials: tomasz konopka, prof, Study Director — Wroclaw Medical University; kamil jurczyszyn, Study Chair — Wroclaw Medical University
Locations (1):
- Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No